CLINICAL TRIAL: NCT02984475
Title: The Potential Hepatoprotective Effect of Metformin in Patients With Beta Thalasemia Major
Brief Title: The Potential Hepatoprotective Effect of Metformin in Patients With Beta Thalassemia Major
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mona Sobhy Abd El-Mon'em Gaber, Teaching assistant-faculty of pharmacy-Cairo University, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CL 1726
Record Dates: First submitted 2016-11-25; First posted 2016-12-07 (Estimated); Last update posted 2018-07-18 (Actual); Status verified 2018-07

CONDITIONS: Beta Thalassemia Major Anemia
Keywords: Beta Thalassemia; Metformin; Oxidative stress; Iron overload; Liver function
MeSH Terms: conditions — beta-Thalassemia; Iron Overload | interventions — Metformin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- treatment arm (Active Comparator): 30 patients receiving blood transfusion and taking iron-chelating therapy along with metformin tablets (500 mg once daily for the first week then twice daily for 6 months).
  Interventions: Drug: Metformin
- control arm (No Intervention): 30 patients receiving blood transfusion and taking iron-chelating therapy.

INTERVENTIONS:
Drug: Metformin
  Other Names: Cidophage
  Arms: treatment arm

SUMMARY:
Beta Thalassemia is a major public health problem in Mediterranean countries.In Egypt, it is considered as the most common chronic hemolytic anemia.one of the major complications in this inherited disorder is iron overload which lead to oxidative stress and tissue damage.

Regarding toxic effect of iron overload on liver, hepatomegaly is one of the most findings that resulting from hemosiderosis, extra medullary hematopoiesis, transmitted hepatitis B and C and cirrhosis.

A lot of studies have been carried out recently to study the beneficial role of metformin in non-diabetic patients of different disorders as non-alcoholic fatty liver disease (NAFLD).Among several studies, it's demonstrated that metformin significantly improved insulin resistance, aminotransferase levels and liver morphology.

The role of metformin in these studies is mainly thought to be antioxidant and anti-inflammatory effects. However, the role of Metformin on hepatic function in different populations with the same mechanism of liver injury should be further investigated.

This clinical trial will be carried out on 60 patients with beta thalassemia major receiving regular blood transfusion and iron chelating therapy, either HCV positive or negative patients.

They will be randomly distributed into either control group (group 1, n=30) receiving blood transfusion and taking iron chelating therapy or treatment group (group 2, n=30) receiving blood transfusion and taking iron chelating therapy along with metformin tablets (500 mg/twice daily) for 6 months.

DETAILED DESCRIPTION:
Beta-Thalassemia is a major public health problem in Mediterranean countries , parts of North and West Africa, the Middle East, the Indian subcontinent, southern Far East and southeastern Asia is of the highest incidence. In Egypt, it is considered as the most common chronic hemolytic anemia (85.1%) with 5.3- 9% carrier rate and annual birth of 1000/1.5 million live births. Thalassemia is a heterogeneous group of hereditary anemia that results from reduced or absent production of alpha or beta globin chains of hemoglobin A. β-thalassemia patients have partial or complete lack of production of β-chains of hemoglobin. The remaining excess of α-chains are unstable, and they finally precipitate and disintegrate, causing red blood cell (RBC) membrane damage. The affected RBCs are prematurely hemolysed in the spleen and bone marrow, leading to increased RBC turnover, ineffective erythropoiesis, and severe anemia that can only be controlled by regular blood transfusion.

One of the major complications in this inherited disorder is iron overload because of premature hemolysis, ineffective erythropoiesis and repeated transfusion in the plasma and major organs such as heart, liver, and endocrine glands. Iron has a catalytic role to produce powerful reactive oxidant species (ROS) and free radicals, which lead to oxidative stress and damage . Children with beta thalassemia have oxidative stress and antioxidant deficiency even without iron overload status. The only way to avoid the accumulation of potentially toxic iron is iron chelation along with the transfusional therapy, desferrioxamine is a chelating agent that has been discovered 30 years ago and since then it has been considered to be one of the most important chelating agent that have been extensively used in the clinical practice . Then other iron chelating agents have been discovered as deferasirox (Exjade®) and deferiprone (Kelfer®). However, there are a lot of problems regarding the compliance to desferrioxamine regimen and the side effects of other orally active iron chelating agents, which rises the need for studying the effect of other naturally occurring iron chelating agents and supplements to reduce the consequences of the iron overload. As reactive oxygen species (ROS) and iron overload have an important role in the pathophysiology of thalassemia , some studies have been carried out to determine the effects of supplements such as silymarin and vitamin E in thalassemic patients on regular blood transfusion and desferrioxamine, and they showing benefit due to their antioxidant, cytoprotective, and iron-chelating activities .

Regarding the toxic effect of iron overload on liver, hepatomegaly is one of the most findings that resulting from hemosiderosis, extra medullary hematopoiesis, transmitted hepatitis B and C and cirrhosis . In one study, liver function tests (LFT) and serum ferritin were elevated in most patients in spite of desferoxamine use .

Metformin (Biguanides) is used as a first-line treatment for patients with type 2 diabetes mellitus . But it is not the only use of metformin, a lot of studies have been carried out recently to study the beneficial role of metformin in non-diabetic patients of different disorders. Metformin was shown to be safe and effective for management of type 2 diabetes in pediatric patients aged 10-16 years old, initiated dose of 500 mg twice daily and titrated up to a maximum of 2000 mg/day based on response . Several clinical studies have supported the beneficial role of metformin in patients with non-alcoholic fatty liver disease (NAFLD) . Most of these studies have evaluated the effect of different doses of metformin on liver biochemistry (aminotransferase profile), histology, and metabolic syndrome feature . Among several studies, it's demonstrated that metformin significantly improved insulin resistance, aminotransferase levels, and liver morphology. Furthermore, in ob/ob mice, a model of hepatic steatosis, it has been shown that metformin reversed hepatomegaly, hepatic fat accumulation, and ALT abnormalities, by reducing hepatic tumor necrosis factor-α (TNF-α) expression . Also the hepatoprotective effect of metformin on methotrexate-induced hepatotoxicity in rabbits with acute lymphocytic leukemia (ALL) has been established. The role of metformin in these studies is mainly thought to be antioxidant and anti-inflammatory effects. However, the role of Metformin on hepatic function in different populations with the same mechanism of liver injury should be further investigated.

This study is conducted to determine the safety and efficacy of metformin as hepatoprotective and antioxidant therapy in iron overloaded patients with Beta-Thalassemia Major.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Beta-Thalassemia Major and receiving regular blood transfusion and on iron chelating therapy.
* Weight: equal to or over 35 kg.
* Normal renal function.

Exclusion Criteria:

* Patients with renal impairment (serum creatinine more than twice the upper limit of normal).
* Patients with heart failure.
* Patients with sepsis or active infection.
* Patients with diabetes mellitus (either primary or secondary to thalassemia).
* regular consumption of medication with potential hepatotoxicity.
* regular herbal medicine or antioxidant supplementation.
* patients with gastrointestinal conditions preventing adsorption of oral medication.

Ages: 11 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-12; Primary Completion 2018-12 (Estimated); Study Completion 2019-04 (Estimated)

PRIMARY OUTCOMES:
liver enzymes tests. | 6 months
  Alanine aminotransferase (ALT) and Aspartate aminotransferase (AST).

SECONDARY OUTCOMES:
Metformin Safety - Number of participants with treatment-related adverse events | 6 months
  Number of participants with treatment-related adverse events as assessed by CTCAE v4.0
liver enzymes and function tests - Alkaline phosphatase (ALP). | 6 months.
  Alkaline phosphatase (ALP).
liver enzymes and function tests - Gama-Glutamyl transferase (GGT). | 6 months.
  Gama-Glutamyl transferase (GGT).
liver enzymes and function tests - total and direct bilirubin. | 6 months.
  total and direct bilirubin.
liver enzymes and function tests - Albumin. | 6 months.
  Albumin .
liver enzymes and function tests - International Normalized Ratio (INR). | 6 months.
  International Normalized Ratio (INR).
oxidative stress markers (MDA). | 6 months.
  Malondialdehyde (MDA)
oxidative stress markers (TAC). | 6 months.
  Total antioxidant capacity (TAC).

OTHER OUTCOMES:
Fibroscan. | 6 months
  Fibroscan will be done for each patient before and at the end of the study.
FIB 4 score. | 6 months
  Fibrosis 4 score.
APRI score. | 6 months
  AST to platelet ratio index score.

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Abo El Reesh Hospital, Cairo
  - El Demerdash (Ain Shams Teaching Hospital)., Cairo